CLINICAL TRIAL: NCT04994769
Title: The Effect of Extended Use of the Epitomee Capsule on Body Weight in Subjects With Overweight and Obesity With and Without Prediabetes
Brief Title: The Effect of Extended Use of the EPITOMEE CAPSULE (ELECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epitomee medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-05-032
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Epitomee Capsule (Experimental): Epitomee Capsule combined with lifestyle counseling
  Interventions: Device: Epitomee Capsule

INTERVENTIONS:
Device: Epitomee Capsule — Epitomee Capsule combined with lifestyle counseling.
  Other Names: The MODEL IBT Program

SUMMARY:
The Effect of Extended Use of the Epitomee Capsule on BodyWeight in subjects with Overweight and Obesity with and without Prediabetes

DETAILED DESCRIPTION:
This is an interventional, open label, single arm extension study to assess the long-term safety and efficacy of the Epitomee Capsule in subjects who completed a 24-week treatment period with the Epitomee-Capsule and experienced at least 3% weight loss during that period. All participating subjects will receive the Epitomee capsule arm in combination with lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Signing an informed consent form prior to any study activity
2. Completed 24 weeks of the core study with maximum of two unattended visits
3. Had at least 3% weight loss in week 24 visit of the core study
4. Non-pregnant, evidenced by a negative urine dipstick pregnancy test by visit 24 week of the core study
5. Females will be either surgically sterile or postmenopausal or agree to continue using an accepted method of birth control during the study
6. Subjects with prediabetes could be untreated or treated with a stable dose of metformin up to 2000 mg/dL inclusive, for at least 1 month prior to entry into the study
7. Currently not using and willingness to avoid non-steroidal anti-inflammatory drugs (NSAIDs) including Diclofenac, Ibuprofen, Naproxen excluding the use of low dose aspirin (75-100 mg) or Celebrex 200-400 mg.
8. Able and willing to continue the lifestyle intervention program as required in the core study including diet and physical activity
9. Subjects must have a primary care physician (PCP) who is responsible for providing routine care
10. Subjects must have cellphone and internet service to communicate with study staff
11. Study subjects must be willing to notify the staff of any change in their medical health (including surgeries) or change in drug treatments (addition of drugs, stopping of drugs, or change in drug dose) during the course of the study
12. Subjects must be willing to avoid medications or other substances known to affect weight changes during the study
13. Subjects on psychiatric medications are clinically well-controlled with a stable psychiatric medication dose for 3 months prior to entry into the extension study

Exclusion Criteria:

1. Currently receiving chronic steroid or immunosuppressive therapy
2. Intending to undergo gastric surgery or gastric banding during the study period.
3. Currently suffering from structural or functional disorders of the esophagus that may impede passage of the device through the gastrointestinal tract, including: Barrett's esophagus, esophagus motility disorder, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation, esophageal motility disorder, esophageal chest pain disorders or any other disorder of the esophagus
4. Currently suffering from swallowing disorder, or drug refractory esophageal reflux symptoms
5. Currently suffering from structural or functional disorders of the stomach including, gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (> 2 cm), cancer or any other disorder of the stomach or any symptoms of chronic upper abdominal pain, chronic nausea, chronic vomiting, chronic dyspepsia or symptoms suggestive of gastroparesis, including post-prandial fullness or pain, post-prandial nausea or vomiting or early satiety.
6. Currently suffering from duodenal ulcer, small bowel diverticula (diverticulitis), intestinal varices, intestinal stricture/stenosis, small bowel obstruction, or any other obstructive disorder of the gastrointestinal (GI) tract
7. Currently having ongoing symptoms suggestive of intermittent small bowel obstruction, such as recurrent bouts of post-prandial abdominal pain, nausea or vomiting
8. Currently having irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease
9. Subjects with Fasting Plasma Glucose ≥126 mg/dL or HbA1c ≥ 6.5% based on blood test results at 24 week visit of the core study
10. Any medications known to be gastric irritants for 4 weeks prior to study start
11. Subjects with congestive heart failure (New York Heart Association (NYHA) Class II, III or IV; myocardial infarction (MI) and/or revascularization (e.g. coronary bypass graft/stent) within 12 months of study start
12. Currently having poorly controlled hypertension (≥ 160 mmHg systolic or ≥ 100 mmHg diastolic)
13. Subjects for whom any anti-platelet drugs beside low dose of Aspirin, have been initiated within 6 months prior to study start
14. Subjects for whom any medications for hypertension or hyperlipidemia have been initiated within 1 month prior to study start
15. Subjects for whom any anti-seizure or anti-arrhythmic medications have been initiated within 6 months prior to study start
16. Subjects who are habitual laxative users or using prescription medication for chronic constipation
17. Any other condition that, in the opinion of the investigator, would interfere with subject participation, may confound the study results, or interfere with compliance with the study (e.g., psychosocial issues, renal disease, hepatic disease, pulmonary disease or cancer disease).
18. Subjects presenting poor abilities and inconsistencies in using the study app during the core study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence, causality, and severity of serious adverse events, potentially related to Epitomee capsule | 24 weeks
  Incidence, causality, and severity of serious adverse events, potentially related to Epitomee capsule during the course of the study
Change in percent weight loss | 24 weeks
  Change in percent weight loss between baseline weight of the Epitomee core study and week 24 of the extension study

SECONDARY OUTCOMES:
Overall incidence, causality and severity of adverse events, potentially related to Epitomee capsule. | 24 weeks
  Overall incidence, causality and severity of adverse events, potentially related to Epitomee capsule during the course of the study
Proportion of subjects who maintain loss of 3% or more of their body weight | 24 weeks
  Proportion of subjects who maintain loss of 3% or more of their body weight from baseline of the Epitomee core study to week 24 of the extension study
Proportion of subjects who lose or maintain loss of 5 % or more of their body weight | 24 weeks
  Proportion of subjects who lose or maintain loss of 5 % or more of their body weight from baseline of the Epitomee core study to week 24 of the extension study
Change in plasma fasting glucose | 24 weeks
  Change in plasma fasting glucose from baseline of the Epitomee core study to week 24 of the extension study
Change in glycemic status (Normoglycemia, Prediabetes and Diabetes) | 24 weeks
  Change in glycemic status (Normoglycemia, Prediabetes and Diabetes) between the Epitomee core study baseline and week 24 of the extension study
Changes in BMI reduction | 24 weeks
  Changes in BMI reduction between baseline BMI in the Epitomee core study and week 24 of the extension study.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Kenan, Dr, Study Director — VP Clinical Affairs
Locations (3):
- United States (3):
  - University of Alabama Department of Nutrition Sciences, Birmingham, Alabama
  - Wake Forest School of Medicine, Wake Forest Baptist Health - 525 Vine Street, 5th Floor, Suite 5119, Winston-Salem, North Carolina
  - Center for Weight and Eating Disorders at Perelman School of Medicine University of Pennsylvania - 3400 Civic Center Boulevard, Building 421,, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Kamar M, Ryan DH, Leonard S, Wyatt HR, Kenan Y, Asaraf LC, Ganon-Elazar E, Ard JD. The safety and efficacy of extended use of an oral shape-shifting superabsorbent hydrogel capsule for weight loss: The ELECT extension study. Obes Pillars. 2025 Oct 20;16:100216. doi: 10.1016/j.obpill.2025.100216. eCollection 2025 Dec. PMID 41216379